CLINICAL TRIAL: NCT01214252
Title: A Retrospective Study Evaluating the Use of Permacol Surgical Implant in the Repair of Abdominal Wall Defects
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVPERH0046
Record Dates: First submitted 2010-09-30; First posted 2010-10-05 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-04

CONDITIONS: Abdominal Wall Defects
Keywords: Repair of patients' abdominal wall defects

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Permacol Patients: Patients who have undergone surgical repair of their abdominal wall defect with Permacol Surgical Implants with at least 12 months follow up.
  Interventions: Device: Permacol Surgical Implant

INTERVENTIONS:
Device: Permacol Surgical Implant — Permacol Surgical Implant

SUMMARY:
To evaluate short, mid and long term clinical outcomes associated with the use of Permacol in the treatment of abdominal wall defects.

ELIGIBILITY:
Inclusion Criteria:

* Equal or over 18 years of age
* Had undergone surgical repair or reconstruction of abdominal wall defects, ventral hernias or incisional hernias using Permacol Surgical Implant.
* At least 12 months of follow-up post date of surgery (-30 days)
* Undergone open or laparoscopic repairs

Exclusion Criteria:

* Had undergone inguinal, parastomal, diaphragmatic or paraesophageal/hiatal hernia repair
* Any prior use of Permacol in abdominal wall repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone surgical repair of their abdominal wall defects with Permacol Surgical Implants with at least 12 months(-30days)follow-up
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Annie Choi, Bedford, Massachusetts, United States

REFERENCES:
- [Derived] Chand B, Indeck M, Needleman B, Finnegan M, Van Sickle KR, Ystgaard B, Gossetti F, Pullan RD, Giordano P, McKinley A. A retrospective study evaluating the use of Permacol surgical implant in incisional and ventral hernia repair. Int J Surg. 2014;12(4):296-303. doi: 10.1016/j.ijsu.2014.01.025. Epub 2014 Feb 5. PMID 24508570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Permacol Patients
Started | 425
Completed | 343
Not Completed | 82
Not completed — Not eligible per protocol | 82

BASELINE CHARACTERISTICS:
Arm/Group | Permacol Patients
Number analyzed (Participants) | 343
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 236
  >=65 years | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 181
Region of Enrollment [Number; unit: participants]
  Europe | 109
  United States | 234

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Hernia Recurrence
Description: Confirmed hernia or hernia recurrence: Proportion of patients treated with Permacol Surgical Implant who experienced hernia or hernia recurrence at the repair site. Hernia or recurrence is defined by hernia diagnosis during clinical assessment by surgeon or medical chart review
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Permacol Patients
Number analyzed (Participants) | 343
participants | 20

2. Secondary Outcome: Total Unconfirmed Hernia or Hernia Recurrence
Description: Total unconfirmed hernia or hernia recurrence at the repair site by year (Number and percentage)
  Unconfirmed hernia or recurrence reported by the subject is defined by confirmation of hernia symptoms based on results of the Symptoms Questionniare but not confirmed by clinical assessment by a surgeon or medical chart review
Time Frame: 12 Months
Measure: Number; unit: participants
Groups:
- Permacol Patients: Total (confirmed or unconfrimed) hernia or hernia recurrence at the repair site by year (# and percentage).
  Unconfirmed hernia or recurrence reported by the subject is defined by confirmation of hernia symptoms based on results of the Symptoms questionnaire but not confirmed by clinical assessment by a surgeon or medical chart review
Arm/Group | Permacol Patients
Number analyzed (Participants) | 343
participants | 9

3. Secondary Outcome: Hernia or Hernia Recurrence by Year From Year 2 to Last Year Observed
Description: Confirmed and Unconfirmed hernia or hernia recurrence by year from Year 2 to last year observed
Time Frame: Year 2 to Year 8
Measure: Number; unit: participants
Arm/Group | Permacol Patients
Number analyzed (Participants) | 343
participants
  Year 2- out of 320 pts | 26
  Year 3- out of 133 pts | 19
  Year 4- out of 67 pts | 5
  Year 5- out of 25 pts | 4
  Year 6- out of 13 pts | 1
  Year 7- out of 6 pts | 1
  Year 8- out of 2 pts | 0

ADVERSE EVENTS:
Description: There were no AEs collected for this study.
Arm/Group | Permacol Patients
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No